CLINICAL TRIAL: NCT03416335
Title: A First-in-Human Phase 1/2 Trial to Determine the Safety and the Pharmacokinetic Profile of DSP-0509, a Synthetic Toll-Like Receptor 7 (TLR-7) Agonist, Administered as Monotherapy and in Combination With Pembrolizumab in Adult Patients With Advanced Solid Tumors
Brief Title: A Study of DSP-0509 in Patients With Advanced Solid Tumors to Determine the Safety and the Pharmacokinetic Profile
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor's decision to terminate the development of the program due to changing landscape.
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BBI-DSP0509-101
Record Dates: First submitted 2018-01-24; First posted 2018-01-31 (Actual); Results first posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Neoplasms
Keywords: DSP-0509; Toll-Like Receptor 7 (TLR-7); BLRM (Bayesian Logistic Regression Model)
MeSH Terms: conditions — Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Monotherapy Arm - Part A (Experimental): Dose Escalation Drug DSP-0509
  Interventions: Drug: DSP-0509
- Combination arm - Part B (Experimental): Dose Escalation Drug DSP-0509, Pembrolizumab
  Interventions: Drug: DSP-0509, Pembrolizumab
- Combination arm - Part C (Experimental): Dose Expansion, Drug DSP-0509, Pembrolizumab
  Interventions: Drug: DSP-0509, Pembrolizumab

INTERVENTIONS:
Drug: DSP-0509 — Each patient treated will receive DSP-0509 at the dose fixed for that Part or cohort administered as a constant rate IV infusion over 10 minutes using a syringe pump.
  Arms: Monotherapy Arm - Part A
Drug: DSP-0509, Pembrolizumab — Each patient treated will receive DSP-0509 at the dose fixed for that Part or cohort administered as a constant rate IV infusion over 10 minutes using a syringe pump and is given in combination with pembrolizumab which should be administered following the dosing schedule of the approved label (200 mg IV q3w)
  Arms: Combination arm - Part B
Drug: DSP-0509, Pembrolizumab — Each patient treated will receive DSP-0509 at the Recommended Phase II Dose (RP2D) level as determined in Part B. It is given as a constant rate IV infusion over 10 minutes using a syringe pump and is given in combination with pembrolizumab which should be administered following the dosing schedule of the approved label (400 mg IV q6w)
  Arms: Combination arm - Part C

SUMMARY:
This is a multi-center, Phase 1 / 2 clinical study for patients with advanced solid tumors. The study consists of 2 treatment arms - a monotherapy arm and a combination arm. The monotherapy arm has 1 part: Dose Escalation (Part A). The combination arm has Dose Escalation (Part B) only.

DETAILED DESCRIPTION:
The primary objective of Monotherapy Arm A is to determine the MTD or RP2D of DSP-0509 when administered as a single agent. Approximately 21 to 30 patients with advanced solid tumors will be enrolled. Several provisional dose levels of DSP-0509, with approximately 3 to 6 patients at each level may be tested in patients with advanced solid tumors. DSP-0509 will be administered as a single agent q2w beginning on Day 1.

The primary objective of Combination Therapy Arm B is to determine the RP2D of DSP-0509 when administered in combination with pembrolizumab, using a BLRM approach. The combination arm will enroll approximately 21 to 30 patients with advanced solid tumors that are (a) metastatic or unresectable and recurrent, and/or refractory to available therapy, (b) a condition for which pembrolizumab is an approved treatment, and (c) in patients who have shown either primary or acquired resistance to an ICI. DSP-0509 will be administered on Day 1 and then every 2 weeks thereafter. Pembrolizumab will be initiated on Day 1.

The primary objective of Combination Therapy Arm C is to determine preliminary efficacy in the form of the ORR of DSP-0509 when administered in combination with pembrolizumab to an expansion cohort of patients with HNSCC, using a Bayesian Adaptive design approach. Combination Arm C will enroll approximately 20 to 40 patients with HNSCC tumors that are (a) metastatic or unresectable, and recurrent and/or refractory to available therapy, (b) in patients who have been treated with pembrolizumab or other PD-1 or PD-L1 inhibitors in monotherapy, and (c) who have subsequently shown either primary or acquired resistance to ICIs.

Dose escalation of DSP-0509 in combination with 400 mg pembrolizumab q6w will start at the same dose of DSP-0509 as the highest (not exceeding the MTD) level tested in the combination regimen with 200 mg pembrolizumab q3w. Upon completion of the DLT evaluation period for the first DSP-0509 dose level tested in combination with 400 mg pembrolizumab q6w in newly enrolled patients, if this dose level is found not to exceed the MTD, any ongoing patients receiving DSP-0509 in combination with pembrolizumab 200 mg q3w will be allowed, at the investigator's discretion, to transition to the 400 mg pembrolizumab q6w regimen, while maintaining the originally assigned DSP-0509 dose level.

ELIGIBILITY:
Inclusion Criteria:

Patients must fulfill each of the following requirements:

1. Must have a histologically or cytologically confirmed advanced solid tumor that meets the following additional specifications

1. Monotherapy Part A (Dose Escalation) advanced solid tumor that is metastatic or unresectable and recurrent and /or refractory to available therapy.
2. Combination Part B (Dose Escalation)- advanced solid tumors that are (a) metastatic or unresectable and recurrent and/or refractory to available therapy; (b) a condition for which pembrolizumab is an approved treatment: and (c) in patients who either have shown primary or acquired resistance to immune checkpoint inhibitors (ICIs)
3. Combination Arm C (Dose Expansion), Phase 2 - Advanced HNSCC tumors of the oropharynx, oral cavity, hypopharynx, larynx, lip, or sinus that are (a) metastatic or unresectable, and recurrent and/or refractory to available therapy, (b) in patients who have been treated with pembrolizumab or other PD-1 or PD-L1 inhibitors in monotherapy, and (c) who have subsequently shown primary or acquired resistance to ICIs.

   For enrollment in both arms:

   2. Must be ≥ 18 years of age

   3. Should have all side effects of any prior therapy or procedures for any medical condition recovered to CTCAE ≤ Grade 1 (except alopecia).

   4. Must have at least 1 measurable lesion by computed tomography or magnetic resonance imaging per RECIST v1.1.

   5. Must have a life expectancy ≥ 3 to 6 months.

   6. Female patients of childbearing age and women < 12 months since the onset of menopause, except those who have been surgically sterilized (tubal ligation) or whose sexual partner(s) is surgically sterilized (vasectomy), must agree to use acceptable contraceptive methods for the duration of the study and for 9 months after the date of their last DSP-0509 infusion. If employing contraception, 2 of the following precautions must be used: birth control pill, vaginal diaphragm, intrauterine system or device, condom or vaginal spermicide. Female patients who are postmenopausal are defined as those with an absence of menses for ≥ 12 consecutive months. Male patients must be surgically sterilized (vasectomy) or their female sexual partner(s) must be surgically sterilized (tubal ligation) to avoid using contraception. If they do not meet this criterion, then male patients or must agree to use a condom as well as one of the acceptable contraceptive methods listed above with their female partner(s) who meets the criteria of either being of childbearing age or is < 12 months since the onset of menopause. Male patients and their female partner(s) must agree to use acceptable contraception methods for the duration of time the male patient is on the study and for 9 months after the date of his last DSP 0509 infusion.

   7. Females of childbearing potential must have a negative serum pregnancy test.

   8. Must have an Eastern Cooperative Oncology Group performance status of 0 to 1.

   9. Must have adequate coagulation function at Screening as determined by:

a. Prothrombin international normalized ratio < 1.5. b. Partial thromboplastin time < 1.5 times the upper limit of normal (ULN).

10. Must have adequate hematologic function at Screening as determined by:

a. White blood cell (WBC) count ≥ 3,000/microliter. b. Absolute neutrophil count (ANC) ≥ 1,500/microliter (patient may not use granulocyte colony stimulating factor or granulocyte-macrophage colony stimulating factor to achieve these WBC and ANC levels).

c. Platelet count ≥ 100 × 103/microliter. d. Hemoglobin (Hgb) ≥ 9.0 g/dL (may not transfuse or use erythropoietin to obtain this Hgb level).

11. Must have adequate renal and hepatic function at Screening as determined by:

1. Serum creatinine < 2.0 mg/dL or < 1.5 times the ULN, whichever is lower.
2. Total bilirubin ≤ 1.5 mg/dL or < 1.5 times the ULN, whichever is lower (or ≤ 2.0 mg/dL for patients with known Gilbert syndrome).
3. Aspartate aminotransferase ≤ 2.5 times ULN (≤ 5 times ULN for patients with liver metastases).
4. Alanine aminotransferase ≤ 2.5 times ULN (≤ 5 times ULN for patients with liver metastases).

   12. Must be able to attend study visits as required by the protocol.

   13. Prior to the first DSP-0509 infusion, the patient must be able to provide tumor tissue for baseline studies either as (a) a block of archival tissue sufficient to provide the required number of slides (b) a sufficient number of fixed, unstained slides of archival tissue or (c) consent to undergo tumor biopsy to acquire sufficient tumor tissue. (Sites need to refer to the current version of the "Sample Collection & Shipment Instructions Manual" to determine how many slides are required for each patient as these numbers vary based on (a) the study Arm/Part in which the patient is enrolled and (b) whether the patient consented to optional future testing).

   In addition to the above criteria, patients must meet the following criteria to be eligible to enroll in Combination Arm C:

   14. Have at least one accessible tumor for biopsy. This accessible lesion must be considered as non-measurable per RECIST criteria, v1.1.

   15. Be platinum refractory, PD-1 or PD-L1 exposed, and have no more than 3 lines of prior therapy for advanced/metastatic disease

   16. Have a known status of PD-L1 combined positive score (CPS)

   17. Have a known HPV status

   Exclusion Criteria:

   Patients with any of the following will be excluded from the study:

   For enrollment in both arms:
   1. Has received prior therapy with a TLR agonist, excluding a topical TLR agonist.
   2. Has received anticancer chemotherapy (including molecular-targeted drugs), radiotherapy, immunotherapy (eg, vaccines or cytokines), or investigational agents within the 3 weeks before the first dose of DSP-0509. Local palliative radiotherapy is permitted3. Receives concurrent systemic (oral or IV) steroid therapy > 10 mg prednisone daily or its equivalent for an underlying condition.

   4. Not fully recovered from major surgery before the first dose of DSP-0509.

   5. Has central nervous system (CNS) metastases (including leptomeningeal metastases, spinal metastases) or CNS primary tumors, eg, glioblastoma.

   6. Has a history of seizures other than isolated febrile seizure in childhood; has a history of a cerebrovascular accident or transient ischemic attack less than 6 months ago.

   7. Has effusions (pleural, pericardial, or ascites) requiring drainage.

   8. Has a neurodegenerative disease, eg, motor neuron disease, Parkinson disease, Alzheimer disease, Huntington disease.

   9. Has retinal detachment, ulcerative keratitis, uveitis, Vogt-Koyanagi-Harada syndrome, choroidal neovascularization, retinopathy/retinitis, thyroid-associated orbitopathy, idiopathic orbital inflammation, diabetic retinopathy, ischemic retinopathy including glaucoma-associated retinopathy, retinal vein thrombosis, or a non-healing ocular or ophthalmic disease.

   10. Has a fever ≥ 38°C within 3 days before the first dose of study treatment.

   11. Has interstitial lung disease or active noninfectious pneumonitis.

   12. Has a history of active autoimmune or immunologic disorder requiring immunosuppression with steroids or other immunosuppressive agents (eg, azathioprine, cyclosporine A) except for patients with isolated vitiligo, resolved childhood asthma or atopic dermatitis, controlled hypoadrenalism or hypopituitarism, and euthyroid patients with a history of Grave disease. Patients with controlled hyperthyroidism must be negative for thyroglobulin, thyroid peroxidase antibodies, and thyroid-stimulating immunoglobulin before study drug administration.

   13. Has a known hypersensitivity to a component of the protocol therapy, DSP-0509, or another pyrimidine.

   14. Has a history of another primary cancer within the 5 years before enrollment except for the following: non-melanoma skin cancer, cervical carcinoma in situ, superficial bladder cancer, or other nonmetastatic carcinoma that has been in complete remission without treatment for more than 5 years.

   15. Has abnormal ECGs that are clinically significant, such as QT prolongation (QTc > 480 msec).

   16. In the opinion of the treating Investigator, has any concurrent conditions that could pose an undue medical hazard or interfere with the interpretation of the study results; these conditions include, but are not limited to ongoing or active infection, clinically significant non-healing or healing wounds, concurrent congestive heart failure (New York Heart Association Functional Classification Class II, III or IV), concurrent unstable angina, concurrent cardiac arrhythmia requiring treatment (excluding asymptomatic atrial fibrillation), recent (within the prior 12 months) myocardial infarction, acute coronary syndrome within the previous 12 months, significant pulmonary disease (shortness of breath at rest or on mild exertion) for example due concurrent severe obstructive pulmonary disease, concurrent hypertension requiring more than 2 medications for adequate control, or diabetes mellitus with more than 2 episodes of ketoacidosis in the prior 12 months.

   17. Has an ejection fraction of 50% or less based on a MUGA scan or ECHO.

   18. Has the presence of a known active acute or chronic infection including human immunodeficiency virus as determined by enzyme-linked immunosorbent assay and confirmed by Western blot; and hepatitis B virus and hepatitis C virus as determined by hepatitis B surface antigen and hepatitis C serology.

   19. Has a cognitive, psychological, or psychosocial impediment that would impair the ability of the patient to receive therapy according to the protocol or adversely affect the ability of the patient to comply with the informed consent process, protocol, or protocol-required visits and procedures.

   20. Receives concurrent strong inhibitors of cytochrome P450 2C8.

   21. Receives concurrent inhibitors of organic anion transporting peptide (OATP)1B1 and OATP1B3.

   22. Is pregnant or breastfeeding.

   23. Has active neurological or inflammatory or auto immune disorders (e.g. Guillain-Barre Syndrome, Amyotrophic Lateral Sclerosis)

   The following exclusion applies only to enrollment in Combination arms Part B & C:

   24. Has a history of immune-related adverse events (irAEs) resulting in permanent discontinuation of ICI treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Indiana University Health Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Henry-Joyce Cancer Center, Vanderbilt University, Nashville, Tennessee
  - M.D. Anderson Cancer Center, The University of Texas, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-six patients were enrolled into the Phase 1 (dose escalation) portion of this study. The study was terminated due to Sponsor's considerations, and therefore the MTD and RP2D have not been determined. No patients were enrolled into the Phase 2 (dose expansion) portion of the study.
Pre-assignment Details: Participants who progressed, died, withdrew consent to survival follow up or were lost to follow up were considered to have completed the study.
Groups:
- Monotherapy Arm - Cohort 1: 0.3mg of DSP-0509 monotherapy administered as an IV constant rate over 3 minutes weekly for 4 weeks followed by biweekly dosing.
- Monotherapy Arm - Cohort 2: 1.0mg of DSP-0509 monotherapy administered as an IV constant rate over 3 minutes weekly for 4 weeks followed by biweekly dosing.
- Monotherapy Arm - Cohort 3: 1.5mg of DSP-0509 monotherapy administered as an IV constant rate over 3 minutes weekly for 4 weeks followed by biweekly dosing.
- Monotherapy Arm - Cohort 4: 1.5mg of DSP-0509 monotherapy administered as an IV constant rate over 10 minutes every 2 weeks.
- Monotherapy Arm - Cohort 5: 2.4mg of DSP-0509 monotherapy administered as an IV constant rate over 10 minutes every 2 weeks.
- Monotherapy Arm - Cohort 6: 3.5mg of DSP-0509 monotherapy administered as an IV constant rate over 10 minutes every 2 weeks.
- Combination Arm - Cohort 1: 0.3mg DSP-0509 administered once weekly, with 200mg pembrolizumab administered once every 3 weeks
- Combination Arm - Cohort 2: 0.3mg DSP-0509 administered twice weekly, with 200mg pembrolizumab administered once every 3 weeks
- Combination Arm - Cohort 3: 1.0mg DSP-0509 administered twice weekly, with 200mg pembrolizumab administered once every 3 weeks
- Combination Arm - Cohort 4: 1.0mg DSP-0509 administered twice weekly, with 400mg pembrolizumab administered once every 6 weeks
Period: Overall Study
Arm/Group | Monotherapy Arm - Cohort 1 | Monotherapy Arm - Cohort 2 | Monotherapy Arm - Cohort 3 | Monotherapy Arm - Cohort 4 | Monotherapy Arm - Cohort 5 | Monotherapy Arm - Cohort 6 | Combination Arm - Cohort 1 | Combination Arm - Cohort 2 | Combination Arm - Cohort 3 | Combination Arm - Cohort 4
Started | 3 | 4 | 5 | 3 | 4 | 7 | 1 | 3 | 3 | 3
Completed | 3 | 4 | 5 | 3 | 4 | 7 | 1 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Monotherapy Arm - Cohort 1 | Monotherapy Arm - Cohort 2 | Monotherapy Arm - Cohort 3 | Monotherapy Arm - Cohort 4 | Monotherapy Arm - Cohort 5 | Monotherapy Arm - Cohort 6 | Combination Arm - Cohort 1 | Combination Arm - Cohort 2 | Combination Arm - Cohort 3 | Combination Arm - Cohort 4 | Total
Number analyzed (Participants) | 3 | 4 | 5 | 3 | 4 | 7 | 1 | 3 | 3 | 3 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 3 | 2 | 2 | 6 | 1 | 1 | 3 | 2 | 26
  >=65 years | 0 | 1 | 2 | 1 | 2 | 1 | 0 | 2 | 0 | 1 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 1 | 2 | 4 | 0 | 2 | 2 | 2 | 16
  Male | 2 | 3 | 4 | 2 | 2 | 3 | 1 | 1 | 1 | 1 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 6
  White | 2 | 3 | 3 | 3 | 4 | 5 | 1 | 2 | 3 | 3 | 29
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLTs) Within the First 6 Weeks of Dosing
Time Frame: From the time of first dose to 6 weeks after the first dose
Measure: Count of Participants; unit: Participants
Arm/Group | Monotherapy Arm - Cohort 1 | Monotherapy Arm - Cohort 2 | Monotherapy Arm - Cohort 3 | Monotherapy Arm - Cohort 4 | Monotherapy Arm - Cohort 5 | Monotherapy Arm - Cohort 6 | Combination Arm - Cohort 1 | Combination Arm - Cohort 2 | Combination Arm - Cohort 3 | Combination Arm - Cohort 4
Number analyzed (Participants) | 3 | 4 | 5 | 3 | 4 | 7 | 1 | 3 | 3 | 3
Participants | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0

2. Primary Outcome: Determination of the Recommended Phase 2 Dose (RP2D) by Assessing Dose-limiting Toxicities (DLTs)
Time Frame: 28 days
Population: Sponsor's decision to terminate the study. Data were not collected to determine the RP2D.
Groups:
- Monotherapy Arm - Part A (Phase I): Dose Escalation DSP-0509 Monotherapy: Each patient received DSP-0509 monotherapy according to dose cohort level administered as a constant rate IV infusion
- Combination Arm - Part B (Phase 1): Dose Escalation Drug DSP-0509 in combination with Pembrolizumab: Each patient received DSP-0509 at the dose fixed for that Part or cohort administered as a constant rate IV infusion over 10 minutes using a syringe pump and is given in combination with pembrolizumab, which should be administered following the dosing schedule of the approved label (200 mg IV every 3 weeks).
Arm/Group | Monotherapy Arm - Part A (Phase I) | Combination Arm - Part B (Phase 1)
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Determination of the MTD of DSP-0509 When Given in Combination With Pembrolizumab by Assessing Dose-limiting Toxicities (DLTs).
Description: MTD of DSP-0509 in patients enrolled into the Combination Arm during the dose escalation part of the study.
Time Frame: 28 days
Population: Sponsor's decision to terminate the study. Data were not collected.
Arm/Group | Combination Arm - Part B (Phase 1)
Number analyzed (Participants) | 0

4. Primary Outcome: Determination of RP2D of DSP-0509 When Given in Combination With Pembrolizumab by Assessing DLTs
Description: Data to be derived from patients enrolled into the Combination Arm - Part B (Phase 1).
Time Frame: 28 days
Population: Sponsor's decision to terminate the study. Data were not collected.
Arm/Group | Combination Arm - Part B (Phase 1)
Number analyzed (Participants) | 0

5. Primary Outcome: Preliminary Antitumor Activity of DSP-0509 in Combination With Pembrolizumab in Patients With Head & Neck Squamous Cell Carcinoma (HNSCC) Who Have Shown Primary or Acquired Resistance to Immune Checkpoint Inhibitors (ICIs)
Description: Data to be derived from patients enrolled into the Combination Arm - Part C (Phase 2)
Time Frame: 4 weeks
Population: Sponsor's decision to terminate study. No patients were enrolled into phase 2 of the study.
Groups:
- Combination Arm - Part C (Phase 2): Dose Expansion Drug DSP-0509 in combination with Pembrolizumab: Each patient received DSP-0509 at the Recommended Phase II Dose (RP2D) level as determined in Part B. It is given as a constant rate IV infusion over 10 minutes using a syringe pump and is given in combination with pembrolizumab, which should be administered following the dosing schedule of the approved label (400 mg IV every 6 weeks)
Arm/Group | Combination Arm - Part C (Phase 2)
Number analyzed (Participants) | 0

6. Secondary Outcome: Evaluate Pharmacokinetics (PK) for Single Agent DSP-0509 by Assessing Plasma Concentration.
Description: Data to be derived from patients enrolled into the Monotherapy Arm - Part A (Phase 1)
Time Frame: 8 weeks
Population: Sponsor's decision to terminate study. Data were not collected.
Groups:
- Monotherapy Arm - Part A (Phase I): Dose Escalation DSP-0509 Monotherapy: Each patient received DSP-0509 monotherapy administered as a constant rate IV infusion over 10 minutes using a syringe pump.
Arm/Group | Monotherapy Arm - Part A (Phase I)
Number analyzed (Participants) | 0

7. Secondary Outcome: Objective Response Rate (ORR) by RECIST
Description: Defined as the proportion of patients with a documented complete response or partial response (CR + PR) based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Time Frame: From date of first dose to 6 months post first dose
Population: Sponsor's decision to terminate study. Data were not collected.
Arm/Group | Monotherapy Arm - Part A (Phase I) | Combination Arm - Part B (Phase 1) | Combination Arm - Part C (Phase 2)
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: ORR by Immune RECIST (iRECIST)
Description: Defined as the proportion of patients with a documented complete response or partial response (CR + PR) based on iRECIST.
Time Frame: From date of first dose to 6 months post first dose
Population: Sponsor's decision to terminate study. Data were not collected.
Arm/Group | Monotherapy Arm - Part A (Phase I) | Combination Arm - Part B (Phase 1) | Combination Arm - Part C (Phase 2)
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Duration of Response (DoR) by RECIST
Description: Defined as the time from first documentation of response until the time of first documentation of disease progression by RECIST v1.1.
Time Frame: 6 months
Population: Sponsor's decision to terminate study. Data were not collected.
Arm/Group | Monotherapy Arm - Part A (Phase I) | Combination Arm - Part B (Phase 1) | Combination Arm - Part C (Phase 2)
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: DoR by iRECIST
Description: Defined as the time from first documentation of response until the time of first documentation of disease progression by iRECIST.
Time Frame: 6 months
Population: Sponsor's decision to terminate study. Data were not collected.
Arm/Group | Monotherapy Arm - Part A (Phase I) | Combination Arm - Part B (Phase 1) | Combination Arm - Part C (Phase 2)
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Progression Free Survival (PFS) by RECIST
Description: Defined as the time from first dose to the earlier date of assessment of progression or death by any cause in the absence of progression by RECIST v1.1.
Time Frame: 12 months
Population: Sponsor's decision to terminate study. Data were not collected.
Arm/Group | Monotherapy Arm - Part A (Phase I) | Combination Arm - Part B (Phase 1) | Combination Arm - Part C (Phase 2)
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: PFS by iRECIST
Description: Defined as the time from first dose to the earlier date of assessment of progression or death by any cause in the absence of progression by iRECIST.
Time Frame: 12 months
Population: Sponsor's decision to terminate study. Data were not collected.
Arm/Group | Monotherapy Arm - Part A (Phase I) | Combination Arm - Part B (Phase 1) | Combination Arm - Part C (Phase 2)
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Evaluate Single Agent DSP-0509-induced Changes in Cytokine Levels.
Description: Data to be derived from patients enrolled into the Monotherapy Arm - Part A (Phase 1)
Time Frame: 8 weeks
Population: Sponsor's decision to terminate study. Data were not collected.
Arm/Group | Monotherapy Arm - Part A (Phase I)
Number analyzed (Participants) | 0

14. Secondary Outcome: Evaluate Change in Cytokine Levels Induced by DSP-0509 in Combination With Pembrolizumab.
Description: Data to be derived from patients enrolled into the Combination Arm - Part B (Phase 1)
Time Frame: 8 weeks
Population: Sponsor's decision to terminate study. Data were not collected.
Arm/Group | Combination Arm - Part B (Phase 1)
Number analyzed (Participants) | 0

15. Secondary Outcome: Evaluate Pharmacokinetics (PK) for Combo Agents DSP-0509 and Pembrolizumab by Assessing Plasma Concentration.
Description: Data to be derived from patients enrolled into the Combination Arm - Part B (Phase 1)
Time Frame: 8 weeks
Population: Sponsor's decision to terminate study. Data were not collected.
Arm/Group | Combination Arm - Part B (Phase 1)
Number analyzed (Participants) | 0

16. Other Pre Specified Outcome: Identification of Potential Metabolites of DSP-0509 in Plasma and Possibly in Urine.
Description: Data to be derived from patients enrolled into the Monotherapy Arm - Part A (Phase 1)
Time Frame: 8 weeks
Population: Sponsor's decision to terminate study. Data were not collected.
Arm/Group | Monotherapy Arm - Part A (Phase I)
Number analyzed (Participants) | 0

17. Other Pre Specified Outcome: Exploratory Pharmacodynamic Evaluation as Potential Biomarkers Capable of Predicting the Clinical Efficacy or Toxicity
Time Frame: 12 months
Population: Sponsor's decision to terminate study. Data were not collected.
Arm/Group | Monotherapy Arm - Part A (Phase I) | Combination Arm - Part B (Phase 1) | Combination Arm - Part C (Phase 2)
Number analyzed (Participants) | 0 | 0 | 0

18. Other Pre Specified Outcome: Exploratory Pharmacodynamic Evaluation as Potential Efficacy-related Immune Response Biomarkers.
Time Frame: 12 months
Population: Sponsor's decision to terminate study. Data were not collected.
Arm/Group | Monotherapy Arm - Part A (Phase I) | Combination Arm - Part B (Phase 1) | Combination Arm - Part C (Phase 2)
Number analyzed (Participants) | 0 | 0 | 0

19. Other Pre Specified Outcome: Evaluate the Effect of DSP-0509 on Cardiac Parameters by Assessing Continuous 25-hour ECG Recordings.
Description: Data to be derived from patients enrolled into Monotherapy Arm - Part A (Phase 1)
Time Frame: 12 months
Population: Sponsor's decision to terminate study. Data were not collected.
Arm/Group | Monotherapy Arm - Part A (Phase I)
Number analyzed (Participants) | 0

20. Other Pre Specified Outcome: Evaluate the PFS Rate as a Potential Evaluation of Treatment Benefit of DSP-0509 Administered With Pembrolizumab
Description: Data to be derived from patients enrolled into Combination Arm - Part C (Phase 2)
Time Frame: 12 months
Population: Sponsor's decision to terminate study. No patients were enrolled into Phase 2 of the study.
Arm/Group | Combination Arm - Part C (Phase 2)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Serious and Other Adverse Events were assessed from the date of first treatment through 30 days of the last administration of study drug, an average of 4 months. All-Cause Mortality was assessed from the date of first treatment until death, an average of 6 months.
Description: Analysis of patients enrolled into each dose cohort during the dose escalation was not done; therefore no data are available for reporting. The outcome reported is based on the totality of AEs and SAEs reported in each arm during phase 1 of the study. No patients were enrolled into phase 2 of the study.
Arm/Group | Monotherapy Arm - Cohort 1 | Monotherapy Arm - Cohort 2 | Monotherapy Arm - Cohort 3 | Monotherapy Arm - Cohort 4 | Monotherapy Arm - Cohort 5 | Monotherapy Arm - Cohort 6 | Combination Arm - Cohort 1 | Combination Arm - Cohort 2 | Combination Arm - Cohort 3 | Combination Arm - Cohort 4
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4 | 1/5 | 0/3 | 1/4 | 1/7 | 0/1 | 0/3 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/4 | 2/5 | 1/3 | 1/4 | 3/7 | 1/1 | 1/3 | 2/3 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 5/5 | 3/3 | 4/4 | 7/7 | 1/1 | 3/3 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Monotherapy Arm - Cohort 1 (N=3) | Monotherapy Arm - Cohort 2 (N=4) | Monotherapy Arm - Cohort 3 (N=5) | Monotherapy Arm - Cohort 4 (N=3) | Monotherapy Arm - Cohort 5 (N=4) | Monotherapy Arm - Cohort 6 (N=7) | Combination Arm - Cohort 1 (N=1) | Combination Arm - Cohort 2 (N=3) | Combination Arm - Cohort 3 (N=3) | Combination Arm - Cohort 4 (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Uveitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Duodenal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cytokine release syndromes (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Encephalitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infections (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Monotherapy Arm - Cohort 1 (N=3) | Monotherapy Arm - Cohort 2 (N=4) | Monotherapy Arm - Cohort 3 (N=5) | Monotherapy Arm - Cohort 4 (N=3) | Monotherapy Arm - Cohort 5 (N=4) | Monotherapy Arm - Cohort 6 (N=7) | Combination Arm - Cohort 1 (N=1) | Combination Arm - Cohort 2 (N=3) | Combination Arm - Cohort 3 (N=3) | Combination Arm - Cohort 4 (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 4 | 1 | 3 | 3 | 0 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Excessive cerumen production (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blurred vision (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Optic nerve disorder (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Trichiasis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Uveitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vitreous detachment (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 3 | 0 | 2 | 2 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 2 | 1 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Duodenal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 1 | 3 | 2 | 3 | 2 | 1 | 1 | 1 | 2
Malaise (General disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Generalized oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Corona virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Encephalitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Onychomycosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Protein urine present (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood calcium increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood phosphorous increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Musculoskeleton pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aura (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine abnormality (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Hot Flush (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
The sponsor made the decision to terminate the study on August 2022 with all patients removed from treatment and follow-up by December 2022. Consistent with Food and Drug Administration and International Council for Harmonisation guidance on the content for abbreviated and synoptic CSRs, only safety data are analyzed and reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-09-15): https://cdn.clinicaltrials.gov/large-docs/35/NCT03416335/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-31): https://cdn.clinicaltrials.gov/large-docs/35/NCT03416335/SAP_001.pdf